CLINICAL TRIAL: NCT02372058
Title: Transcutaneous Bilirubinometry in Neonates With Bilicare System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gerium Medical (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 10002
Record Dates: First submitted 2015-02-22; First posted 2015-02-26 (Estimated); Results first posted 2015-09-11 (Estimated); Last update posted 2015-09-11 (Estimated); Status verified 2015-08

CONDITIONS: We Will Focus on Assessing the Clinical Performance of the BiliCare Device

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BiliCare (Other): Three non invasive measurements of TcB:
  Two measurements with the BiliCare device and one measurement with a competitive FDA approved device
  Interventions: Device: BiliCare

INTERVENTIONS:
Device: BiliCare — Three non invasive measurements of TcB:
  Two measurements with the BiliCare device and one measurement with a competitive FDA approved device

SUMMARY:
The primary objective of this study is to define the performance evaluation of BiliCare TcB device to the "gold standard" bilirubin tests.

DETAILED DESCRIPTION:
Neonatal hyperbilirubinemia or newborn jaundice impacts over 85% of all newborns [1]. Regardless of the mechanism, excessive hyperbilirubinemia has been traditionally treated with phototherapy to minimize any probable risk of developing bilirubin-induced neurotoxicity. However, earlier and more recent data suggest that pre-discharge bilirubin screening for risk of significant hyperbilirubinemia, whether due to a rapid bilirubin production or an earlier age of onset, has impacted the guidelines for clinical use of phototherapy [1, 2]. In this study, we plan to test the performance of a novel transcutaneous device (BiliCareTM) first for screening for bilirubin levels at postnatal age of 6 to 48 hrs; and possibly also, to substitute the use of this measurement for total plasma/serum bilirubin (TB). This device applies a novel light transmission technology that has the potential to measure bilirubin as a point-of-care test in the subcutaneous tissue, and then uses an internal algorithm to calculate bilirubin levels in the skin. In this proposalstudy, we will to assess the clinical performance of the BiliCare by correlating measurements made by this device to near-concurrent measure of total plasma/serum bilirubin at normative ranges (mean, median, range and inter-quartile ranges ) for all term and late-preterm newborns (including those who are at-risk for jaundice and / or being administered with phototherapy) born to families of diverse race and ethnic backgrounds.

ELIGIBILITY:
Inclusion Criteria:

* Parental informed consent
* Male and female newborns with a GA ≥ 35 wks
* Enrollment at age > 6 hrs until neonatal discharge.
* Pre-phototherapy

Exclusion Criteria:

* Infants requiring respiratory assistance (such as mechanical ventilation)
* Severe or life-threatening congenital anomalies
* Hematomas at the point of measurement on both ears
* Neonates undergone blood transfusion

Min Age: 6 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2014-09; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Schutzman, MD, Principal Investigator — Einstein Medical Center
Locations (1):
- Einstein Medical Center, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Late Preterm and Term Newborns: The study population will consist of term and late preterm newborns (infants >=35 weeks gestational age)
Period: Overall Study
Arm/Group | Late Preterm and Term Newborns
Started | 103
Completed | 100
Not Completed | 3
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Population: Number of participants who completed the study
Arm/Group | Late Preterm and Term Newborns
Number analyzed (Participants) | 100
Age, Continuous [Mean (Standard Deviation); unit: Hours since birth] | 43.5 (19.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57
  Male | 43
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 23
  Not Hispanic or Latino | 75
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 49
  White | 14
  More than one race | 0
  Unknown or Not Reported | 33

OUTCOME MEASURES:

1. Primary Outcome: BiliCare TcB Result Compared to TSB Result
Time Frame: 30 minutes within taking the blood draw for TSB (either before or after the blood draw)
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- BiliCare TcB Average: The study population will consist of term and late preterm newborns (infants >=35 weeks gestational age) measured with one BiliCare TcB device without an infection control tip and with one BiliCare TcB device with an infection control tip.
  This is the average of both devices
- JM103 TcB: The study population will consist of term and late preterm newborns (infants >=35 weeks gestational age) measured with the JM103 TcB device
- Total Serum Bilirubin (TSB): The study population will consist of term and late preterm newborns (infants >=35 weeks gestational age) measured routinely for total serum bilirubin by diazo method.
Arm/Group | BiliCare TcB Average | JM103 TcB | Total Serum Bilirubin (TSB)
Number analyzed (Participants) | 100 | 100 | 100
mg/dL | 8.46 (2.68) | 7.93 (3.48) | 7.83 (3.27)

ADVERSE EVENTS:
Arm/Group | Late Preterm and Term Newborns
Serious Adverse Events (participants affected / at risk) | 0/100
Other Adverse Events (participants affected / at risk) | 0/100

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No